CLINICAL TRIAL: NCT05227469
Title: The Effect of Myofunctional Exercises in Class II Patients
Brief Title: Myofunctional Therapy Twin Block
Acronym: twin block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BezmialemVU myofunctional
Record Dates: First submitted 2022-01-12; First posted 2022-02-07 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Malocclusion, Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Myofunctional Therapy

STUDY DESIGN:
Intervention Model Description: Double blinded controlled clinical study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the care provider will know which patients had only twin block treatment and which patients had both twin block and egzersize treatment. Control group will have unrevealant egzercises or no egzercises.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skeletal class II twinblock + myofunctional therapy (Experimental): Myofunctional exercises will be prescribed in addition to the standart twin block therapy. Movements will be taught to this group, for which we have prescribed the exercises. It will be ensured that the exercises are done more properly and regularly by taking video recordings every other day from the group that does the exercises twice a day. Incorrect exercises will be corrected by providing feedback.
  Interventions: Behavioral: myofunctional therapy
- Control (No Intervention): Standard twin block therapy will be used for Class II patients. Patients will be informed that they are involved in a study that follows growth and development, and they will receive feedback on whether they use their devices properly, but no myofunctional exercise.

INTERVENTIONS:
Behavioral: myofunctional therapy — In order to confirm that the exercises are done for a sufficient time and are done correctly, the researcher will take video recordings from the participants and examine these recordings every other day. Respondents will be contacted when errors are detected.
  Arms: Skeletal class II twinblock + myofunctional therapy

SUMMARY:
There are situations where orthodontic treatment cannot provide long-term benefits. The proposed orthotropic theory proposes that environmental factors cause malocclusion and genes decide its pattern. The primary aim of this project is to increase the success, aesthetics and permanence of the treatment result by providing the best facial change of the pediatric patients in the MP3cap period, and that myofunctional exercises can be used in addition to orthodontic treatments during the treatment process of the patients.

DETAILED DESCRIPTION:
Many studies in recent years have emphasized the importance of the environmental factor as well as the hereditary causes of malocclusion. In particular, the activity and posture of the oral soft tissues have begun to be mentioned more. In the presence of bad habits, there are cases where orthodontic treatment alone is not sufficient and must be combined with myofunctional treatments. There are also many physicians who emphasize the importance of positioning the tongue in contact with the palate during swallowing and resting.

It is known that habits during growth and development cause malocclusions that may occur in the future. It may be possible to acquire some myofunctional exercises as a habit during the growth and development period as a prophylactic solution against malocclusions. In addition to twin block treatment, myofunctional exercises will be given to class II pediatric patients in the MP3cap period, and the effect of exercises on oral soft and hard tissues will be compared at the end of the treatment. The effects of tongue and lip movements on facial development as well as on the treatment process will be examined. Perhaps in the future, everyone can recommend doing myofunctional exercises in addition to tooth brushing.

ELIGIBILITY:
Inclusion Criteria:

1. Having a skeletal Class II relationship (ANB > 4°),
2. Skeletal Class II relationship due to mandibular retrognathia (SNB < 78°),
3. Overjet is more than 5 mm,
4. Normal growth pattern SN-GoGn (32° ± 6°),
5. Minimum crowding of the dental arch is 4 mm or less,
6. Bilateral Class II molar and canine relationship is at least 3.5 mm,
7. Patients who are in MP3 cap period will be taken according to the Tanner-Whitehouse wrist and wrist X-ray method.

Exclusion Criteria:

1. Having received orthodontic treatment before,
2. Having severe maxillary stenosis,
3. Severe facial asymmetry according to clinical and x-ray analysis,
4. Poor oral hygiene,
5. Having mental retardation at a level that will affect the patient's cooperation,

7. Having a systemic disease that will affect the orthodontic treatment, 8. Congenital anomaly or syndrome.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
SNB Angle (sella-nasion-point B Angle at cephalometric analysis) | 6 months
  Cephalometric analysis can be performed to evaluate the cranial base, the relationship of the maxilla to the cranial base, the mandible's size and position relative to the cranial base, the relationship between the maxilla and the mandible, the vertical dimension, maxillary and mandibular dentition, and soft tissue. The angle between the sella/nasion plane and nasion/B plane (normal value at the end of growth 80 ± 2°). This angle assesses the antero-posterior position of the mandible relative to the upper cranial structures. SNB indicates whether or not the mandible is normal, prognathic, or retrognathic.
SNA Angle (sella-nasion-point A Angle at cephalometric analysis) | 12 months
  Cephalometric analysis can be performed to evaluate the cranial base, the relationship of the maxilla to the cranial base, the mandible's size and position relative to the cranial base, the relationship between the maxilla and the mandible, the vertical dimension, maxillary and mandibular dentition, and soft tissue. SNA is the the angle between the sella/nasion plane and the nasion/A plane (normal value at the end of growth 82 ± 2°). This angle assesses the antero-posterior position of the maxilla relative to the upper cranial structures. It indicates whether or not the maxilla is normal, prognathic, or retrognathic.
ANB Angle (point A-nasion-point B Angle at cephalometric analysis) | 12 months
  The difference between SNA and SNB angles
PASmin mm (PAS min = The shortest distance between base of the tongue and the posterior wall of the pharynx at cephalometric analysis) | 12 months
  The minimal distance between the base of the tongue and the posterior pharyngeal wall, representing the minimal pharyngeal airway space

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kılıç, asst. prof, Study Director — Bezmialem Vakıf Üniversitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Banu Kilic, Istanbul, Fatih
  - Banu Kılıç, Fatih, Istanbul

IPD SHARING:
Plan to Share IPD: No